CLINICAL TRIAL: NCT00003385
Title: A Phase I Study of Paclitaxel, Carboplatin, and Increasing Doses of Doxil in Untreated Ovarian, Peritoneal, and Tubal Carcinoma
Brief Title: Combination Chemotherapy in Treating Patients With Untreated Ovarian, Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000066381; GOG-9703
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2003-09

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; ovarian undifferentiated adenocarcinoma; ovarian mixed epithelial carcinoma; ovarian serous cystadenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian clear cell cystadenocarcinoma; fallopian tube cancer; primary peritoneal cavity cancer; Brenner tumor
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Brenner Tumor | interventions — Carboplatin; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy consisting of liposomal doxorubicin, paclitaxel, and carboplatin in treating patients who have untreated ovarian, peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of doxorubicin HCl liposome when administered with paclitaxel and carboplatin in patients with previously untreated ovarian epithelial, peritoneal, or fallopian tube cancer.
* Determine the toxicity of this treatment regimen in these patients.
* Evaluate measurable disease in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of doxorubicin HCl liposome (LipoDox).

Patients receive LipoDox IV on day 1, carboplatin IV over 3 hours on days 1 and 22, and paclitaxel IV over 1 hour on days 1, 8, 15, 22, 29, and 36. Treatment repeats every 42 days for 4 courses in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of LipoDox until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. An additional cohort of 12 patients receives LipoDox at the MTD with carboplatin and paclitaxel as above.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 48 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed previously untreated ovarian epithelial carcinoma, peritoneal carcinoma, or fallopian tube carcinoma
* The following histologic epithelial cell types are eligible:

  * Serous adenocarcinoma
  * Endometrioid adenocarcinoma
  * Mucinous adenocarcinoma
  * Undifferentiated carcinoma
  * Clear cell adenocarcinoma
  * Mixed epithelial carcinoma
  * Transitional cell
  * Malignant Brenner tumor
  * Adenocarcinoma not otherwise specified
* No more than 12 weeks since diagnosis
* No ovarian epithelial carcinoma of low malignant potential (borderline carcinomas)

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Absolute granulocyte count at least 1,500/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times normal
* SGOT/SGPT no greater than 3 times normal
* Alkaline phosphatase no greater than 3 times normal
* Gamma-glutamyl-transferase no greater than 3 times normal
* No acute hepatitis

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance greater than 50 mL/min

Cardiovascular:

* LVEF normal by MUGA
* No unstable angina
* No myocardial infarction within the past 6 months
* Patients with abnormal cardiac conduction (e.g., bundle branch block or heart block) are eligible if disease has been stable for the past 6 months

Other:

* No septicemia or severe infection
* No severe gastrointestinal bleeding
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* Recovered from recent prior surgery

Other:

* No prior anticancer therapy that would preclude study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 1999-03; Primary Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter G. Rose, MD, Study Chair — MetroHealth Cancer Care Center at MetroHealth Medical Center
Locations (8):
- United States (7):
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - University of Texas Medical Branch, Galveston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Norwegian Radium Hospital, Oslo, Norway

REFERENCES:
- [Result] Rose PG, Greer BE, Horowitz IR, Markman M, Fusco N. Paclitaxel, carboplatin and pegylated liposomal doxorubicin in ovarian and peritoneal carcinoma: a phase I study of the Gynecologic Oncology Group. Gynecol Oncol. 2007 Jan;104(1):114-9. doi: 10.1016/j.ygyno.2006.07.036. Epub 2006 Sep 7. PMID 16959305
- [Result] Rose PG, Greer BE, Markman M, et al.: A phase I study of paclitaxel, carboplatin, and liposomal doxorubicin in ovarian, peritoneal, and tubal carcinoma: a Gynecologic Oncology Group Study. [Abstract] Proceedings of the American Society of Clinical Oncology 19: A-1531, 2000.